CLINICAL TRIAL: NCT04169997
Title: A Phase III Study to Evaluate the Efficacy and Safety of IMP4297 Following 1st Line Chemotherapy in the Monotherapy Maintenance Treatment of Subjects With Ovarian Cancer
Brief Title: A Study of IMP4297 as Maintenance Treatment Following First-line Chemotherapy in Patients With Advanced Ovarian Cancer
Acronym: FLAMES
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMP4297-301
Record Dates: First submitted 2019-11-17; First posted 2019-11-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMP4297 (Experimental): The starting dose is 100mg QD
  Interventions: Drug: IMP4927
- Placebos (Placebo Comparator): The starting dose is 100mg QD
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: IMP4927 — IMP4297 tablet.The starting dose from 100mg QD
  Arms: IMP4297
Drug: Placebos — Placebos tablet.The starting dose from 100mg QD
  Arms: Placebos

SUMMARY:
IMP4297 is a PARP inhibitor. This is a 2:1 randomized, double-blind, placebo-controlled study conducted in patients with advanced (FIGO Stage III or IV) ovarian cancer to evaluate Efficacy and Safety of IMP4297 for Maintenance Treatment

DETAILED DESCRIPTION:
A Phase III Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of IMP4297 Following First-Line Platinum-based Chemotherapy in the Monotherapy Maintenance Treatment . The Subjects with newly diagnosed, histologically confirmed FIGO stage lll-IV high grade serous, high grade endometrioid or BRCA mutant other histological types of epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer who have had a complete/partial response (CR/PR) after first-line platinum-based therapy will be randomly assigned to IMP4297 or placebo at a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have the ability to read, communicate effectively with the investigator and sign the ICF in writing. Subjects have to provide ICF prior to any study-specified procedures
* Subjects must be ≥ 18 years of age
* Newly diagnosed, histologically confirmed FIGO stage III-IV high grade serous, high grade endometrioid or BRCA mutant other histological types of epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer (according to local pathological diagnosis) (with concrete staging criteria of FIGO provided in Appendix 7)
* Subjects who have completed first-line platinum-based (carboplatin or cisplatin) chemotherapy (intravenous or intraperitoneal) prior to randomization
* The test results of CA125 before treatment must meet the following specific criteria:
* If the first test value is ≤upper limit of normal (ULN), the subject can be randomized without second sampling
* If the first test value is >ULN, a second assessment must be performed at least 7 days after the first. If the value of the subject's second assessment is ≥15% higher than that of the first, the subject is not eligible for inclusion
* Subjects must have normal organ and bone marrow function, as defined below, within 28 days prior to the first dose of investigational drug (corrective treatment with blood products ≤28 days prior to the first dose of investigational drug, such as blood transfusion, is not allowed)
* Eastern Cooperative Oncology Group (ECOG) Performance Status score 0-1
* Subjects must have a life expectancy ≥16 weeks

Exclusion Criteria:

* Participation in the planning and/or conduct of the study (applicable to sponsor staff and/or site staff)

  -BRCA mutation status is unclear
* Subjects with early disease (FIGO stage I or II)

  -Subjects with tumor assessment of SD or PD after first-line chemotherapy
* More than one cytoreductive surgery prior to study randomization. (Subjects with tumor considered unresectable in diagnosis and with biopsy or oophorectomy only, followed by continued chemotherapy and intermittent cytoreductive surgery can be enrolled in the study)
* Subjects with previously diagnosed with early stage ovarian, fallopian tube, or primary peritoneal cancer followed by treatment
* Subjects with previously received chemotherapy for any abdominal or pelvic tumor, including treatment of previously diagnosed early stage ovarian, fallopian tube, or primary peritoneal cancer

  -Subjects with ascites drawn during the last two chemotherapy cycles prior to study enrollment
* Have been randomized in this study
* Have participated in another investigational drug trial during chemotherapy prior to randomization
* History of other malignancies within the past 5 years, except for the following: adequately treated thyroid cancer, non-melanoma skin cancer, effectively treated carcinoma in situ of the cervix, Stage I ductal carcinoma in situ (DCIS), stage I grade 1 endometrial cancer or other solid tumors, including lymphomas (without bone marrow involvement) that have been treated effectively and without evidence of disease for more than 5 years
* Classification II or above severe congestive heart failure assessed by New York Heart Association (NYHA); history of myocardial infarction or unstable angina within 6 months before treatment; history of stroke or transient ischemic attack within 6 months before treatment

  * Any systemic chemotherapy or radiotherapy (except for palliative reasons) within 4 weeks (or longer, depending on the characteristics of the drug used) prior to the first dose of investigational drug
  * Subjects who have received strong CYP3A4 inhibitors or strong CYP3A4 inducers before the first dose of the investigational drug (≥ 5 half-lives of washout period from the first dose of the investigational drug can be enrolled) and need to continue to receive these drugs during the study
* Toxicity from prior anti-tumor therapy has not recovered to ≤ Grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03, except alopecia
* Subjects with myelodysplastic Syndrome (MDS) /Acute Myeloid (AML) Leukemia

  * Have active or untreated metastases in central nervous system; subjects with treated brain metastases can be enrolled if the following criteria is met
  * Have no imaging progression ≥ 4 weeks after the end of treatment (EOT);
  * The treatment completed ≥ 28 days prior to the first dose of investigational drug;
  * Treatment with systemic corticosteroids (> 10 mg/day prednisone or equivalent) is not required ≤ 14 days prior to the first dose of investigational drug
* Have received drugs targeting poly-ADP-ribose polymerase (PARP)

  * Have clinically significant active infection at the discretion of the investigator
  * History of clinically significant liver disease at the discretion of the investigator, including active viral or other hepatitis, history of alcohol abuse, or cirrhosis; except for subjects with previous viral hepatitis confirmed to be inactive by polymerase chain reaction (PCR) assay
  * Have infection of human immunodeficiency virus (HIV)
* Subjects who are unable to swallow oral preparations and with gastrointestinal disorders, so the absorption of the investigational drug may be interfered
* Nursing women
* Subjects with known hypersensitivity to the investigational drug or its excipients
* Have had major surgery within 4 weeks prior to the first dose of investigational drug -Subjects, at the discretion of the investigator, with poor compliance or with any factors unsuitable for participation in this trial; subjects, at the discretion of the investigator, to be unsuitable for participation in this study due to any clinical or laboratory abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 404 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Approximately 42 months since the first subject enrolled
  BICR-assessed progression-free survival (PFS)

SECONDARY OUTCOMES:
CFI | Approximately 42 months since the first subject enrolled
  chemotherapy- free interval assessed by Investigators
PFS2 | Approximately 42 months since the first subject enrolled
  progression-free survival 2 (PFS2) assessed by Investigators
TFST | Approximately 42 months since the first subject enrolled
  Time to first subsequent anti-tumor treatment (TFST)
TDT | Approximately 42 months since the first subject enrolled
  time from randomization to study treatment discontinuation or death (TDT)
os | Approximately 42 months since the first subject enrolled
  the time from the date of randomization to the date of death caused by any reason

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua wu, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu X, Liu J, Wang J, Wang L, Lin Z, Wang X, Zhu J, Kong B, Fei J, Tang Y, Xia B, Liang Z, Wang K, Huang Y, Zheng H, Lin A, Jiang K, Wang W, Wang X, Lou G, Pan H, Yao S, Li G, Hao M, Cai Y, Chen X, Yang Z, Chen Y, Wen H, Qu P, Xu C, Hsieh CY; FLAMES Investigators. Senaparib as first-line maintenance therapy in advanced ovarian cancer: a randomized phase 3 trial. Nat Med. 2024 Jun;30(6):1612-1621. doi: 10.1038/s41591-024-03003-9. Epub 2024 May 15. PMID 38750351